CLINICAL TRIAL: NCT00854776
Title: The Occurrence of Peptic Ulcer Disease and Its Complications in Ischemic Heart Patients Taking Aspirin and Clopidogrel With or Without Co-prescription of Proton Pump Inhibitor
Brief Title: Peptic Ulcer Disease in Ischemic Heart Patients Taking Aspirin and Clopidogrel With or Without Proton Pump Inhibitor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Luo, Jiing-Chyuan, M.D. (Attending Physician of Section of Gastroenterology), Taipei Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V98C1-051
Record Dates: First submitted 2009-03-01; First posted 2009-03-03 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Peptic Ulcer; Ulcer Complications
Keywords: aspirin; clopidogrel; proton pump inhibitor; peptic ulcer; ulcer complications
MeSH Terms: conditions — Peptic Ulcer | interventions — Lansoprazole; Aluminum Hydroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Upper GI tract symptoms are evaluated. Patients are asked to report to gastroenterologist if they have persistent ulcer symptoms and to report to the emergency room if they have evidence of GI bleeding or ulcer complications (melena, hematemesis, or sudden onset of severe epigastric pain). Endoscopy will be undergone to document any gastroduodenal ulcers with or without ulcer complications. If the hemoglobin level has decreased by 2g/dL or more, or stool check shows occult blood at each visit, endoscopy will be undergone to check the presence of gastroduodenal ulcers with or without bleeding. Patients without persistent ulcer symptoms or without evidence of ulcer complications will be invited to undergone scheduled endoscopy at the 3-month end of follow-up in each subjective.
  Interventions: Drug: lansoprazole
- 2 (Placebo Comparator): Upper GI tract symptoms are evaluated at each visit. Patients are asked to report to gastroenterologist if they have persistent ulcer symptoms and to report to the emergency room if they have evidence of GI bleeding or ulcer complications (melena, hematemesis, or sudden onset of severe epigastric pain). Endoscopy will be undergone to document any gastroduodenal ulcers with or without ulcer complications. An ulcer is defined as a circumscribed mucosal break at least 3 mm in diameter. If the hemoglobin level has decreased by 2g/dL or more, or stool check shows occult blood at each visit, endoscopy will be undergone to check the presence of gastroduodenal ulcers with or without bleeding. Patients without persistent ulcer symptoms or without evidence of ulcer complications will be invited to undergone scheduled endoscopy at the 3-month end of follow-up in each subjective.
  Interventions: Drug: aluminum hydroxide 334 mg and Mg hydroxide 166 mg

INTERVENTIONS:
Drug: lansoprazole — 30 mg once daily
  Other Names: Takepron
  Arms: 1
Drug: aluminum hydroxide 334 mg and Mg hydroxide 166 mg — 1 tablet once daily
  Arms: 2

SUMMARY:
Studies showed that combined use of clopidogrel and aspirin had a 25 % reduction of risk on myocardial infarction and stroke in patients who undergone percutaneous coronary intervention (PCI) when compared with use of aspirin alone. However, major GI bleeding rose in combined group than aspirin group. Use of proton pump inhibitor (PPI) which diminishes gastric acid secretion effectively reduces aspirin or clopidogrel associated ulcer or/and ulcer bleeding in general population and high risk patients. The investigator hypothesis is whether use of PPI can reduce ulcer and ulcer complication in patients taking both clopidogrel and aspirin.

DETAILED DESCRIPTION:
Patients are eligible if they have received PCI for their stenotic coronary arteries. Patients who had a past history of PUD without complication, who have taken aspirin or clopidogrel before enrolling for their CV disease will be allowed to enroll. Patients are excluded if they have New York Heart Association class IV heart failure, if they had contraindications to antithrombotic or antiplatelet therapy, if they have clinical severe thrombocytopenia (platelet count< 80000/mm3), if they have previous disabling, or hemorrhagic stroke or intracranial hemorrhage, if they have severe and unstable conditions in hepatic, renal, and pulmonary disease, if they have unstable and progressive malignancy, if they have epigastralgia or have a positive occult blood in stool, if they have current or recent peptic ulcer disease and take PPI or histamine receptor-2 antagonist without proving healed ulcer by scopy, if they have received a surgical intervention due to ulcer complication (bleeding, perforation, obstruction) in the past. Patient will be randomly assigned aspirin (100 mg/day) plus clopidogrel (75 mg/day) with PPI (lansoprazole-Takepron@ 30 mg/day) or aspirin (100 mg/day) plus clopidogrel (75 mg/day) with placebo (antacid 1 table/day) for 3 months. Patients will be followed as outpatients, with visit every one month, checking blood hemoglobin as well as stool occult blood for 3 months.Patients are asked to report to gastroenterologist if they have persistent ulcer symptoms (epigastric pain, dyspepsia) and to report to the emergency room if they have evidence of GI bleeding or ulcer complications (melena, hematemesis, or sudden onset of severe epigastric pain). Endoscopy will be undergone to document any gastroduodenal ulcers with or without ulcer complications. Patients without persistent ulcer symptoms or without evidence of ulcer complications will be invited to undergone scheduled endoscopy at the 3-month end of follow-up.The primary end point is the occurrence of clinical upper GI events (symptomatic ulcer and ulcer complications-bleeding, perforation, or obstruction). The secondary end point is occurrence of dyspepsia, asymptomatic gastroduodenal ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if they have received PCI for their stenotic coronary arteries and taken both aspirin and clopidogrel.
* Patients who had a past history of PUD without complication, who have taken aspirin or clopidogrel before enrolling for their CV disease will be allowed to enroll.

Exclusion Criteria:

* Patients are excluded if they have New York Heart Association class IV heart failure, if they had contraindications to antithrombotic or antiplatelet therapy, if they have clinical severe thrombocytopenia (platelet count< 80000/mm3), if they have previous disabling, or hemorrhagic stroke or intracranial hemorrhage, if they have severe and unstable conditions in hepatic, renal, and pulmonary disease, if they have unstable and progressive malignancy, if they have epigastralgia or have a positive occult blood in stool, if they have current or recent PUD and take PPI or histamine receptor-2 antagonist without proving healed ulcer by scopy, if they have received a surgical intervention due to PUD complication (bleeding, perforation, obstruction) in the past, if they have received a GP IIb/IIIa inhibitor fewer than 3 days before randomization.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The primary end point is the occurrence of clinical upper GI events (symptomatic ulcer and ulcer complications-bleeding, perforation, or obstruction) | 3 month follow-up

SECONDARY OUTCOMES:
The secondary end point is occurrence of dyspepsia, asymptomatic gastroduodenal ulcers | 3 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan